CLINICAL TRIAL: NCT00549718
Title: A Phase 3 Randomized, Placebo-Controlled, CLinical Trial to Study the Safety and Efficacy of Three Doses of Lurasidone HCl in Acutely Psychotic Patients With Schizophrenia
Brief Title: Lurasidone HCl: A Phase 3 Study of Patients With Acute Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1050229; 2007-003819-31 (EudraCT Number)
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; SM-13496; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lurasidone 40mg (Experimental)
  Interventions: Drug: Lurasidone HCl
- Lurasidone 80mg (Experimental)
  Interventions: Drug: Lurasidone HCl
- Lurasidone 120mg (Experimental)
  Interventions: Drug: Lurasidone HCl
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: Lurasidone HCl — Once daily

SUMMARY:
Lurasidone HCl is a compound being developed for the treatment of schizophrenia. This clinical study is designed to test the hypothesis that lurasidone is more efficacious than placebo. The study will also evaluate the safety and tolerability of lurasidone as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to enter the study, each patient must comply with the following inclusion criteria:

* Provide written informed consent and aged between 18 and 75 years of age.
* Meets DSM-IV™ criteria for a primary diagnosis of schizophrenia.
* Not pregnant, if of reproductive potential agrees to remain abstinent or use adequate and reliable contraception for duration of study.
* Able and agrees to remain off prior antipsychotic medication for the duration of study.
* Good physical health on the basis of medical history, physical examination, and laboratory screening.
* Willing and able to comply with the protocol, including the inpatient requirements and outpatient visits.

Exclusion Criteria:

* Considered by the investigator to be at imminent risk of suicide or injury to self, others, or property.
* Any chronic organic disease of the CNS (other than schizophrenia)
* Used investigational compound within 30 days.
* Clinically significant or history of alcohol abuse/alcoholism or drug abuse/dependence within the last 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (48):
- United States (21):
  - K&S Professional Research Services, LLC., Little Rock, Arkansas
  - Comprehensive Neuroscience, Inc, Cerritos, California
  - Clinical Innovations, Inc., Costa Mesa, California
  - Collaborative Neuroscience Network Inc.,12772 Valley View Street,Suite 3, Garden Grove, California
  - California Clinical Trials, Paramount, California
  - Pasadena Research Institute, Pasadena, California
  - California Neuropsychopharmacology,CNRI - Los Angeles LLC,8309 Telegraph Road, Pico Rivera, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Comprehensive Neuroscience, Inc., Washington D.C., District of Columbia
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Segal Institute for Clinical Research, Fidelity Clinical Research, Inc., North Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Alexian Brothers Health System, Hoffman Estates, Illinois
  - Lake Charles Clinical Trials LLC, Lake Charles, Louisiana
  - Booker, J. Gary, MD. APMC, Shreveport, Louisiana
  - Center for Behavioral Health, LLC, Rockville, Maryland
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Erie County Medical Center, Corp, Buffalo, New York
  - CRI Worldwide LLC at Kirkbride, Philadelphia, Pennsylvania
  - Research Strategies of Memphis, LLC., Memphis, Tennessee
  - Future Search Trials of Neurology, Austin, Texas
- Hospital Caremeau, Nîmes, France
- India (6):
  - S V Medical College, Tirupati, Andh Prad
  - Government Hospital for Mental Care, Visakhapatnam, Andh Prad
  - Sheth Vadilal Sarabhai General Hospital, Ahmedabad, Gujarat
  - Shanti Nursing Home, Aurangabad, Mahara
  - Madras Medical College & Government General Hospital, Chennai, Tamil Nadu
  - Deva Mental Health Care, Varanasi, Uttar Prad
- Malaysia (2):
  - Hospital Permai, Johor Bahru, Johor
  - University Malaya Medical Centre, Kuala Lumpur
- Romania (5):
  - Spitalul Clinic Judetean de Urgenta Arad, Arad
  - Spitalul de Psihiatrie Titan "Dr. Constantin Gorgos", Bucharest
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia, Bucharest
  - Centrul de Recuperare si Reabilitare Gura Ocnitei, Gura Ocniței
  - Spitalul Judetean Arges, Piteşti
- Russia (7):
  - North State Medical University, Arkhangelsk
  - Republic Psychiatric Hospital, Karelia
  - City Psychoneurological Dispensary #7 (with Hospital), Saint Petersburg
  - City Psyhiatric Hospital #2 of St. Nikolay Chudotvorets, Saint Petersburg
  - City Psychiatric Hospital #4, Saint Petersburg
  - Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - City Psychiatric Hospital #3 of Skvortsov-Stepanov, Saint Petersburg
- Ukraine (6):
  - Dnipropetrovsk Regional Clinical Hospital named Mechnikov, Dnipropetrovsk
  - Reg. Clin. Psychiatric Hosp. DSMU n.af.M.Gorkiy, Donetsk
  - Kyiv City Clin. Psychoneurolog. Hosp.#1, Kyiv
  - Lv. St. Med. Univ. n. af. D. Halytskiy Oblast Clin. Psychon. Hosp, Lviv
  - Odesa SMU, based on Odessa Reg. Psychiatric Hosp.#1, Odesa
  - Kherson Regional Psychiatric Hospital, Vil. Stepanovka, Kherson

REFERENCES:
- [Result] Nasrallah HA, Silva R, Phillips D, Cucchiaro J, Hsu J, Xu J, Loebel A. Lurasidone for the treatment of acutely psychotic patients with schizophrenia: a 6-week, randomized, placebo-controlled study. J Psychiatr Res. 2013 May;47(5):670-7. doi: 10.1016/j.jpsychires.2013.01.020. Epub 2013 Feb 17. PMID 23421963
- [Derived] Hopkins SC, Tomioka S, Ogirala A, Loebel A, Koblan KS, Marder SR. Assessment of Negative Symptoms in Clinical Trials of Acute Schizophrenia: Test of a Novel Enrichment Strategy. Schizophr Bull Open. 2022 Apr 7;3(1):sgac027. doi: 10.1093/schizbullopen/sgac027. eCollection 2022 Jan. PMID 39144777
- [Derived] Hopkins SC, Ogirala A, Worden M, Koblan KS. Depicting Safety Profile of TAAR1 Agonist Ulotaront Relative to Reactions Anticipated for a Dopamine D2-Based Pharmacological Class in FAERS. Clin Drug Investig. 2021 Dec;41(12):1067-1073. doi: 10.1007/s40261-021-01094-7. Epub 2021 Nov 9. PMID 34751928
- [Derived] Correll CU, Cucchiaro J, Silva R, Hsu J, Pikalov A, Loebel A. Long-term safety and effectiveness of lurasidone in schizophrenia: a 22-month, open-label extension study. CNS Spectr. 2016 Oct;21(5):393-402. doi: 10.1017/S1092852915000917. Epub 2016 Apr 6. PMID 27048911
- [Derived] Nasrallah HA, Cucchiaro JB, Mao Y, Pikalov AA, Loebel AD. Lurasidone for the treatment of depressive symptoms in schizophrenia: analysis of 4 pooled, 6-week, placebo-controlled studies. CNS Spectr. 2015 Apr;20(2):140-7. doi: 10.1017/S1092852914000285. Epub 2014 Jun 23. PMID 24955752

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone 40mg: Lurasidone 40 mg tablets taken once a day The number of subjects in the participant flow (overall study) is based on the total number of subjects randomized (500). The number of subjects in the baseline characteristics is based on the safety population (489). All randomized subjects who received at least one dose of study medication were included in the safety analysis. This means that 3 subjects were randomized but never received a dose of study drug.
- Lurasidone 80mg: lurasidone 40m mg tablets taken once/day The number of subjects in the participant flow (overall study) is based on the total number of subjects randomized (500). The number of subjects in the baseline characteristics is based on the safety population (489). All randomized subjects who received at least one dose of study medication were included in the safety analysis. This means that 4 subjects were randomized but never received a dose of study drug.
- Lurasidone 120mg: Lurasidone 40 mg tablets taken once/day
- Placebo: Matching placebo to Lurasidone 40 mg taken once/day The number of subjects in the participant flow (overall study) is based on the total number of subjects randomized (500). The number of subjects in the baseline characteristics is based on the safety population (489). All randomized subjects who received at least one dose of study medication were included in the safety analysis. This means that 4 subjects were randomized but never received a dose of study drug.
Period: Overall Study
Arm/Group | Lurasidone 40mg | Lurasidone 80mg | Lurasidone 120mg | Placebo
Started | 125 | 123 | 124 | 128
Completed | 84 | 86 | 85 | 73
Not Completed | 41 | 37 | 39 | 55
Not completed — Insufficient clinical response | 20 | 7 | 18 | 32
Not completed — Adverse Event | 6 | 8 | 7 | 3
Not completed — Lost to Follow-up | 4 | 2 | 0 | 6
Not completed — Withdrawal by Subject | 9 | 18 | 12 | 13
Not completed — Administrative | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 40mg | Lurasidone 80mg | Lurasidone 120mg | Placebo | Total
Number analyzed (Participants) | 122 | 119 | 124 | 124 | 489
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.1) | 38.6 (9.5) | 37.7 (11.2) | 38.2 (9.9) | 38.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 32 | 34 | 149
  Male | 82 | 76 | 92 | 90 | 340
Region of Enrollment [Number; unit: participants]
  France | 0 | 1 | 1 | 1 | 3
  United States | 70 | 64 | 70 | 67 | 271
  Malaysia | 2 | 2 | 2 | 2 | 8
  Ukraine | 13 | 12 | 12 | 14 | 51
  Romania | 9 | 9 | 9 | 9 | 36
  Russian Federation | 14 | 15 | 13 | 15 | 57
  India | 14 | 16 | 17 | 16 | 63

OUTCOME MEASURES:

1. Secondary Outcome: CGI-S From Baseline to the End of the Double-blind Treatment
Description: Clinical Global Impression of Severity is a clinician-rated assessment of the subject's current illness state on a 7 point scale, where a higher score is associated with greater illness severity. The scale has a single item measured on a 7 point scale from 1 ('normal', not ill) to 7 (extremely ill).
Time Frame: 6 weeks
Population: The primary population for the efficacy analysis was the Intent-to-Treat (ITT) population.All subjects who were randomized, received at least one dose of study medication, and have a Baseline efficacy measurement and at least one post-Baseline efficacy measurement,were in the efficacy analysis in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Lurasidone 40mg | Lurasidone 80mg | Lurasidone 120mg | Placebo
Number analyzed (Participants) | 122 | 119 | 124 | 124
scores on a scale | -1.1 [-1.3 to -0.9] | -1.4 [-1.6 to -1.2] | -1.2 [-1.4 to -1.0] | -1.0 [-1.2 to -0.8]
Statistical Analysis 1: Comparison: Lurasidone 40mg vs Lurasidone 80mg vs Lurasidone 120mg vs Placebo; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Change in Total PANSS Score From Baseline to the End of the Double Blind Phase
Description: The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
Time Frame: 6 weeks
Population: The primary population for the efficacy analysis was the Intent-to-Treat (ITT) population. All subjects who were randomized, received at least one dose of study medication, and have a Baseline efficacy measurement and at least one post-Baseline efficacy measurement, were in the efficacy analysis in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Lurasidone 40mg | Lurasidone 80mg | Lurasidone 120mg | Placebo
Number analyzed (Participants) | 121 | 118 | 123 | 124
scores on a scale | -19.2 [-22.6 to -15.7] | -23.4 [-26.9 to -19.9] | -20.5 [-24.0 to -17.1] | -17.0 [-20.5 to -13.6]
Statistical Analysis 1: Comparison: Lurasidone 40mg vs Lurasidone 80mg vs Lurasidone 120mg vs Placebo; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 14 days post study therapy
Arm/Group | Lurasidone 40mg | Lurasidone 80mg | Lurasidone 120mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/124 | 3/121 | 6/124 | 5/127
Other Adverse Events (participants affected / at risk) | 96/124 | 90/121 | 106/124 | 85/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lurasidone 40mg (N=124) | Lurasidone 80mg (N=121) | Lurasidone 120mg (N=124) | Placebo (N=127)
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 1
Complex Partial Seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Psychotic Disorders (Psychiatric disorders) | 0 | 1 | 1 | 3
Schizophrenia (Psychiatric disorders) | 1 | 1 | 5 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lurasidone 40mg (N=124) | Lurasidone 80mg (N=121) | Lurasidone 120mg (N=124) | Placebo (N=127)
Dyspepsia (Gastrointestinal disorders) | 6 | 7 | 12 | 6
Nausea (Gastrointestinal disorders) | 14 | 8 | 15 | 9
Vomiting (Gastrointestinal disorders) | 5 | 7 | 12 | 5
Weight Increase (Investigations) | 6 | 4 | 9 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 2 | 2
Akathisia (Nervous system disorders) | 14 | 21 | 30 | 65
Dystonia (Nervous system disorders) | 6 | 9 | 3 | 1
Headache (Nervous system disorders) | 23 | 16 | 21 | 20
Parkinsonism (Nervous system disorders) | 8 | 5 | 12 | 0
Sedation (Nervous system disorders) | 7 | 13 | 13 | 6
Somnolence (Nervous system disorders) | 13 | 12 | 18 | 7
Agitation (Psychiatric disorders) | 7 | 3 | 7 | 2
Insomnia (Psychiatric disorders) | 8 | 9 | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multi-center studies, it is mandatory that the first publication is based on all data obtained from all analyses as stipulated in the protocol. Investigators participating in multicenter studies must agree not to present data gathered individually or by subgroup of centers before the full, initial publication, unless this has been agreed to by all other investigators and also by DSP-Sepracor.